CLINICAL TRIAL: NCT03892707
Title: Observational Study of Effectiveness and Safety of Add-on Milgamma® and Milgamma® Compositum Step-Therapy in Routine Practice of Management of Adult Patients With Acute Non-Specific Low Back Pain Receiving Modern NSAIDs
Brief Title: Milgamma® and Milgamma® Compositum Step-therapy in Patients With Acute Non-specific Low Back Pain Receiving Modern NSAID
Status: Completed | Type: Observational
Sponsor: Woerwag Pharma LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: WP-RU-2018/1
Record Dates: First submitted 2019-03-21; First posted 2019-03-27 (Actual); Results first posted 2021-08-27 (Actual); Last update posted 2021-10-06 (Actual); Status verified 2021-09

CONDITIONS: Acute Non-specific Low Back Pain
Keywords: Low back pain; Milgamma; NSAIDs
MeSH Terms: conditions — Low Back Pain | interventions — Celecoxib; Etoricoxib; Meloxicam; nimesulide

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (2):
- NSAIDs group: Patients with acute non-specific low back pain prescribed with modern NSAIDs (preferential/selective COX-2 inhibitors)
- NSAIDs+Milgamma+Milgamma compositum group: Patients with acute non-specific low back pain prescribed with modern NSAIDs (preferential/selective COX-2 inhibitors) + Milgamma® / Milgamma® compositum
  Interventions: Drug: Exposure of interest (within routine clinical practice):Vitamin B complexes Milgamma® and Milgamma® compositum

INTERVENTIONS:
Drug: Exposure of interest (within routine clinical practice):Vitamin B complexes Milgamma® and Milgamma® compositum — Milgamma®: 2 mL injection solution containing thiamin hydrochloride 100 mg, pyridoxine hydrochloride 100 mg, cyanocobalamin 1 mg, lidocaine hydrochloride 20 mg.
  Milgamma® compositum: 1 tablet containing benfotiamine 100 mg, pyridoxine hydrochloride 100 mg.
  Other Names: Non-Steroidal Anti-Inflammatory Drugs (celecoxib, etoricoxib, meloxicam, nimesulide)
  Groups: NSAIDs+Milgamma+Milgamma compositum group

SUMMARY:
The purpose of this study is to assess the effectiveness and safety of add-on Milgamma®/ Milgamma® compositum step-therapy in patients with acute non-specific low back pain receiving modern NSAIDs in routine medical practice.

DETAILED DESCRIPTION:
This is a multi-centre observational prospective study that was planned for assessment the effectiveness of neurotropic vitamins therapy with Milgamma®/ Milgamma® compositum in combination with modern NSAIDs (preferential/selective cyclooxygenase-2 (COX-2) inhibitors) in patients with acute non-specific back pain. Approximately 500 adult out-patients with acute non-specific low back pain who have been prescribed therapy consisting of (1) modern NSAIDs (preferential/selective COX-2 inhibitors) or (2) modern NSAIDs (preferential/selective COX-2 inhibitors) + Milgamma® / Milgamma® compositum will be enrolled in the study. Each patient will be observed over a period of approximately 94 days. 9 visits/phone contacts are planned to be conducted during this period. Information about patient's condition, pain intensity, pain flare-ups, satisfaction with the treatment, patient's disability, therapy used for acute back pain treatment, data on safety will be collected during these contacts. Pain intensity will be measured with Numeric Rating Scale (NRS), patients' disability will be evaluated with Roland Morris disability questionnaire, patients' satisfaction with the treatment will be assessed with 5-point verbal rating scale. Safety assessment will be based on frequency and severity of adverse drug reactions recorded during the study.

Prior to the start of the study, neurologists (potential investigators) will be asked to fill out feasibility questionnaires to identify their individual routine practice regarding prescription or non-prescription of Milgamma® / Milgamma® compositum. Based on results of feasibility physicians will be divided to non-prescribers and prescribers of Milgamma® / Milgamma® compositum to the patients with acute non-specific low back pain. In each medical institution, such non-prescribers and prescribers will be proposed to participate in the study. Non-prescribers will be responsible for enrolling group (1) (NSAIDs alone), prescribers will be responsible for enrolling group (2) (NSAIDs + Milgamma® / Milgamma® compositum).

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent including data protection declaration according to the local legislation.
* Acute non-specific low back pain less than 21 days (= 3 weeks).
* Low back pain treatment with (1) modern NSAIDs (preferential/selective COX-2 inhibitors) or (2) modern NSAIDs (preferential/selective COX-2 inhibitors) + Milgamma®/ Milgamma® compositum prescribed (but not started yet) in frames of routine medical practice.
* Prescribed (but not started yet) step-therapy with Milgamma® to be followed by Milgamma® compositum in accordance with locally approved instruction for medical use (for the group planned to be treated with Milgamma®/ Milgamma® compositum step-therapy).
* Pain intensity according to Numerical Rating Scale (NRS) ≥4 points ≤9 at the time of enrollment.
* In case of presence of previous episodes of acute non-specific low back pain in medical history, the last one had resolved at least 30 days before the start of current episode.

Exclusion Criteria:

* History or presence of any disease that, in the opinion of the investigator, might confound the results of the study, poses an additional risk to the subject during participation in the study or can change pain perception (examples of such possible conditions: any malignancy, stomach ulcer, duodenal ulcer, chronic heart failure, bronchial asthma, psychiatry disorders, epilepsy, Parkinson Disease etc).
* Spinal surgery/rehabilitation in the last 12 months.
* Acute back pain that is attributable to any known or suspected specific identifiable cause (e.g. discogenic radiculopathy, spondylolisthesis, osteomalacia, inflammatory arthritis, metabolic, neurological diseases or tumor).
* Severe scoliosis.
* Use of NSAIDs or vitamins B within 2 months prior to enrollment into the study.
* Necessity to use myorelaxants or antidepressants for treatment of acute non-specific low back pain.
* Prior use of non-pharmacological treatment (physiotherapy, heat treatment (e.g. heat patch, hot water bottle) or topically applied medicinal products to the back area, procaine blocks) within the last 3 days before study entry.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Adult out-patients will be enrolled by neurologists in clinical sites all over the Russian Federation.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2018-12-15 (Actual); Primary Completion 2019-11-05 (Actual); Study Completion 2019-11-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vladimir Parfenov, Study Chair — I.M. Sechenov First Moscow State Medical University
Locations (21):
- Russia (21):
  - LLC Medical Center "Nebolit", Mytishchi, Moscow Oblast
  - LLC "Research Medical Complex "Vashe Zdorovie", Kazan'
  - State Healthcare Institution "Republican Clinical Neurological Center", Kazan'
  - Regional State Budgetary Institution of Health "Regional Clinical Hospital № 1" named after Prof. S.I. Sergeev, Khabarovsk
  - Federal State Healthcare Institution "Russian Scientific Center of Surgery named after academician B.V. Petrovsky", Moscow
  - LLC "Medicina", Moscow
  - Non-state Healthcare Institution "Central Clinical Hospital No. 2 named after N.A. Semashko of the JSC Russian Railways, Moscow
  - LLC "Clinical Diagnostic Center Avitsena", Naberezhnye Chelny
  - LLC "Licon Plus", Naberezhnye Chelny
  - LLC "Medis", Nizhny Novgorod
  - JSC "MEdical Center Avitsenna", group of companies "Mother and Child", Novosibirsk
  - LLC "MRI-Expert Novosibirsk", Novosibirsk
  - LLC "Multidisciplinary center of modern medicine "Euromed", Omsk
  - Federal State Healthcare Institution St. Petersburg Clinical Hospital of the Russian Academy of Sciences, Saint Petersburg
  - Out-patient clinic of SUE St. Petersburg Metropoliten, Saint Petersburg
  - LLC "MD Project 2010", Ufa
  - LLC "National Medical Holding Medstandart", Ufa
  - Volgograd State Medical University, Volgograd
  - LLC "Center of Evidence-Based Medicine", Yaroslavl
  - State Healthcare Institution of Yaroslavl Region "Clinical Hospital №8", Yaroslavl
  - LLC "Center for Medical Prevention and Rehabilitation treatment "Kamkor", Yekaterinburg

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 500 patients with acute non-specific low back pain were enrolled in the study at 56 clinical sites.
Groups:
- NSAIDs Group: Patients with acute non-specific low back pain prescribed with modern NSAIDs (preferential/selective cyclooxygenase-2 (COX-2) inhibitors)
- NSAIDs+Milgamma+Milgamma Compositum Group: Patients with acute non-specific low back pain prescribed with modern NSAIDs (preferential/selective cyclooxygenase-2 (COX-2) inhibitors) + Milgamma® / Milgamma® compositum Milgamma®: 2 mL injection solution containing thiamin hydrochloride 100 mg, pyridoxine hydrochloride 100 mg, cyanocobalamin 1 mg, lidocaine hydrochloride 20 mg.
  Milgamma® compositum: 1 tablet containing benfotiamine 100 mg, pyridoxine hydrochloride 100 mg.
Period: Overall Study
Arm/Group | NSAIDs Group | NSAIDs+Milgamma+Milgamma Compositum Group
Started | 250 | 250
Started Study Treatment at Baseline | 244 | 250
Completed | 244 | 244
Not Completed | 6 | 6
Not completed — Screen failure | 6 | 0
Not completed — Pain resolution | 0 | 4
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Other (long business trip) | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- NSAIDs+Milgamma+Milgamma Compositum Group: Patients with acute non-specific low back pain prescribed with modern NSAIDs (preferential/selective COX-2 inhibitors) + Milgamma® / Milgamma® compositum Milgamma®: 2 mL injection solution containing thiamin hydrochloride 100 mg, pyridoxine hydrochloride 100 mg, cyanocobalamin 1 mg, lidocaine hydrochloride 20 mg.
  Milgamma® compositum: 1 tablet containing benfotiamine 100 mg, pyridoxine hydrochloride 100 mg.
- Total: Total of all reporting groups
Arm/Group | NSAIDs Group | NSAIDs+Milgamma+Milgamma Compositum Group | Total
Number analyzed (Participants) | 244 | 250 | 494
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 244 | 250 | 494
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.6 (10.1) | 42.1 (10.3) | 40.9 (10.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 143 | 142 | 285
  Male | 101 | 108 | 209
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants] — All study participants were enrolled in clinical sites located in different regions of Russian Federation.
  participants
    Russia | 244 | 250 | 494
Pain intensity and patients' disability at baseline [Mean (Standard Deviation); unit: units on a scale] — Pain intensity was measured using 0-10 point Numeric Rating Scale (NRS). NRS is 11-step scale for assessment of pain intensity at the moment of patient's examination ranging from 0 (no pain) to 10 (worst pain imaginable).
  Patients' disability was assessed using Roland Morris disability questionnaire (RMDQ). RMDQ is a 24-item self-administered disability measure in which greater level of pain-related disability is reflected by higher score. The RMDQ score ranges from 0 to 24 with a lower score indicating better function.
  units on a scale
    Pain intensity at baseline | 6.6 (1.2) | 6.7 (1.1) | 6.6 (1.2)
    Patients' disability at baseline | 11.1 (4.8) | 11.7 (4.4) | 11.4 (4.6)

OUTCOME MEASURES:

1. Primary Outcome: Change of Pain Intensity After 10 Days of Treatment
Description: Pain intensity was measured using 0-10 point Numeric Rating Scale (NRS). NRS is 11-step scale for assessment of pain intensity at the moment of patient's examination ranging from 0 (no pain) to 10 (worst pain imaginable). Pain intensity was measured at baseline and at 10 days after the start of treatment.
Time Frame: Baseline; Visit 3 (10 days after the start of treatment)
Population: Full Analysis Set (FAS)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | NSAIDs Group | NSAIDs+Milgamma+Milgamma Compositum Group
Number analyzed (Participants) | 244 | 250
units on a scale | -5.1 (1.8) | -4.0 (1.7)
Statistical Analysis 1: Comparison: NSAIDs Group vs NSAIDs+Milgamma+Milgamma Compositum Group; Since the superiority of one treatment over the other is investigated and taking into consideration that smaller negative values of the primary variable correspond to the greater reduction of pain, the statistical hypotheses are: Null hypothesis (H0): H0: μ2 - μ1 ≥ 0 Alternative hypothesis (HA): HA: μ2 - μ1 < 0, where μ1 и μ2 are the mean changes from baseline in pain intensity for (1) modern NSAIDs therapy and for (2) modern NSAIDs + Milgamma\ Milgamma compositum therapy, correspondingly; Test type: Superiority — The between-group comparison on primary endpoint - change from baseline in pain intensity as measured on 0-10 points NRS scale at 10 days after the start of treatment was performed using analysis of covariance (ANCOVA). The difference between pain intensity at 10 days after the start of treatment and baseline (V3-V1) as response variable, treatment group as fixed factor and baseline pain intensity as a covariate was included into the model; p < 0.001, ANCOVA

2. Secondary Outcome: Change of Pain Intensity After 5, 24 and 38 Days of Treatment
Description: Pain intensity was measured using 0-10 point Numeric Rating Scale (NRS). NRS is 11-step scale for assessment of pain intensity at the moment of patient's examination ranging from 0 (no pain) to 10 (worst pain imaginable). Pain intensity was measured at baseline, at 5, 24 and 38 days after the start of treatment.Changes of pain intensity from baseline to Day 5, from baseline to Day 24 and from baseline to Day 38 after the start of treatment were calculated separately.
Time Frame: Baseline; Visit 2 (5 days after the start of treatment), Visit 4 (24 days after the start of treatment); Visit 5 (38 days after the start of treatment)
Population: Full Analysis Set (FAS)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | NSAIDs Group | NSAIDs+Milgamma+Milgamma Compositum Group
Number analyzed (Participants) | 244 | 250
units on a scale
  Change of pain intensity from baseline to Day 5 after the start of treatment | -3.1 (1.5) | -2.4 (1.3)
  Change of pain intensity from baseline to Day 24 after the start of treatment | -6.1 (1.5) | -5.3 (1.8)
  Change of pain intensity from baseline to Day 38 after the start of treatment | -6.3 (1.4) | -6.0 (1.7)
Statistical Analysis 1: Comparison: NSAIDs Group vs NSAIDs+Milgamma+Milgamma Compositum Group; Changes from baseline in pain intensity measured on 0-10 points NRS scale at 5, 24 and 38 days after were compared between groups using ANCOVA models similar to those used for the analysis of the primary variable; Test type: Superiority; p < 0.001, ANCOVA

3. Secondary Outcome: Change of Pain Intensity Over Time
Description: Pain intensity was measured using 0-10 point Numeric Rating Scale (NRS). NRS is 11-step scale for assessment of pain intensity at the moment of patient's examination ranging from 0 (no pain) to 10 (worst pain imaginable). Pain intensity was measured at baseline, at 5, 10, 24 and 38 days after the start of treatment. A mixed model repeated measures was used to analyze change from baseline in pain intensity over time from Baseline to Visit 5 (38 days after the start of treatment) in each group. The model included a random effect for subject and fixed effect terms for treatment, visit, treatment-by-visit interaction, baseline pain intensity. An unstructured covariance structure was used to model the within-subject errors. P-value was calculated for the difference between treatment groups.
Time Frame: From Baseline to Visit 5 (38 days after the start of treatment)
Population: Full Analysis Set (FAS)
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | NSAIDs Group | NSAIDs+Milgamma+Milgamma Compositum Group
Number analyzed (Participants) | 244 | 250
units on a scale | -5.1 [-5.2 to -4.9] | -4.4 [-4.5 to -4.2]
Statistical Analysis 1: Comparison: NSAIDs Group vs NSAIDs+Milgamma+Milgamma Compositum Group; Test type: Superiority; p < 0.001, ANCOVA

4. Secondary Outcome: Percentage of Patients With 30% Low Back Pain Relief After 5, 10, 24 and 38 Days of Treatment.
Description: Pain intensity was measured using 0-10 point Numeric Rating Scale (NRS). NRS is 11-step scale for assessment of pain intensity at the moment of patient's examination ranging from 0 (no pain) to 10 (worst pain imaginable). Relief in pain intensity was defined as 100%*(pain intensity at baseline - pain intensity at Visit 2, 3, 4 or 5)/ pain intensity at baseline. Percentage of patients showing at least 30% low back pain relief at Visit 2 (5 days after the start of treatment), at Visit 3 (10 days after the start of treatment), at Visit 4 (24 days after the start of treatment) and at Visit 5 (38 days after the start of treatment) were calculated separately.
Time Frame: Visit 2 (5 days after the start of treatment); Visit 3 (10 days after the start of treatment); Visit 4 (24 days after the start of treatment) and Visit 5 (38 days after the start of treatment)
Population: Full Analysis Set (FAS)
Measure: Count of Participants; unit: Participants
Arm/Group | NSAIDs Group | NSAIDs+Milgamma+Milgamma Compositum Group
Number analyzed (Participants) | 244 | 250
Participants
  Number and percentage of patients with 30% pain relief at Day 5 after the start of treatment | 194 | 140
  Number and percentage of patients with 30% pain relief at Day 10 after the start of treatment | 235 | 214
  Number and percentage of patients with 30% pain relief at Day 24 after the start of treatment | 241 | 240
  Number and percentage of patients with 30% pain relief at Day 38 after the start of treatment | 244 | 241
Statistical Analysis 1: Comparison: NSAIDs Group vs NSAIDs+Milgamma+Milgamma Compositum Group; For Visit 2 (5 days after the start of treatment) relief in pain intensity was defined as 100%*(pain intensity at baseline - pain intensity at Visit 2)/ pain intensity at baseline. The denominator for the proportion of patients was the number of patients with available pain intensity measurements after imputation using Last observation carried forward (LOCF) method; Test type: Superiority — Between-group comparison was carried out using logistic regression with treatment group as fixed factor and baseline pain intensity as a covariate. Treatment effect was tested using the corresponding p-value; p < 0.001, Regression, Logistic
Statistical Analysis 2: Comparison: NSAIDs Group vs NSAIDs+Milgamma+Milgamma Compositum Group; For Visit 3 (10 days after the start of treatment) relief in pain intensity was defined as 100%*(pain intensity at baseline - pain intensity at Visit 3)/ pain intensity at baseline. The denominator for the proportion of patients was the number of patients with available pain intensity measurements after imputation using Last observation carried forward (LOCF) method; Test type: Superiority — [test comment as in outcome 4, analysis 1]; p < 0.001, Regression, Logistic
Statistical Analysis 3: Comparison: NSAIDs Group vs NSAIDs+Milgamma+Milgamma Compositum Group; For Visit 4 (24 days after the start of treatment) relief in pain intensity was defined as 100%*(pain intensity at baseline - pain intensity at Visit 4)/ pain intensity at baseline. The denominator for the proportion of patients was the number of patients with available pain intensity measurements after imputation using Last observation carried forward (LOCF) method; Test type: Superiority — [test comment as in outcome 4, analysis 1]; p = 0.061, Regression, Logistic

5. Secondary Outcome: Change in Pain-related Disability After 10 Days of Treatment
Description: Patients' disability was assessed using Roland Morris disability questionnaire (RMDQ). RMDQ is a 24-item self-administered disability measure in which greater level of pain-related disability is reflected by higher score. The RMDQ score ranges from 0 to 24 with a lower score indicating better function.
Time Frame: Baseline; Visit 3 (10 days after the start of treatment)
Population: FAS population
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | NSAIDs Group | NSAIDs+Milgamma+Milgamma Compositum Group
Number analyzed (Participants) | 244 | 250
units on a scale | -8.4 (4.6) | -7.0 (4.0)
Statistical Analysis 1: Comparison: NSAIDs Group vs NSAIDs+Milgamma+Milgamma Compositum Group; Change from baseline in pain-related disability as measured by Roland Morris disability questionnaire at 10 days after the start of treatment was compared between groups using analysis of covariance (ANCOVA) model with treatment group as fixed factor and baseline value disability score as a covariate; Test type: Superiority; p < 0.001, ANCOVA

6. Secondary Outcome: Percentage of Patients With at Least One Pain Flare-up During the Study
Description: Episode of pain flare-up was defined as presence of at least 1 day with low back pain following a period without pain lasting at least 4 weeks. Therefore pain flare-ups were registered no earlier than 4 weeks after the start of treatment, i.e. starting from Visit 5 (38 days after the start of treatment). The occurrence of pain flare-up was determined by the investigator.
Time Frame: From Visit 5 (38 days after the start of treatment) to Visit 9 (End of Study Visit, 94 days after the start of treatment)
Population: Full Analysis Set (FAS). Denominator of proportion was the number of FAS patients who had at least one pain-free period during the study.
Measure: Count of Participants; unit: Participants
Arm/Group | NSAIDs Group | NSAIDs+Milgamma+Milgamma Compositum Group
Number analyzed (Participants) | 240 | 238
Participants | 35 | 10
Statistical Analysis 1: Comparison: NSAIDs Group vs NSAIDs+Milgamma+Milgamma Compositum Group; Episode of pain flare-up was defined as presence of at least 1 day with pain following a period without pain lasting at least 4 weeks . The denominator for the proportion was the number of FAS patients who had at least one pain-free period with approximately 4 weeks duration registered during the study; Test type: Superiority; p < 0.001, Fisher Exact

7. Secondary Outcome: Percentage of Patients With at Least One Pain Flare-up Resulting in Consultancy With Physician, Resulting in Disruption of Daily Activity, and Resulting in NSAIDs Intake
Description: Episode of pain flare-up was defined as presence of at least 1 day with low back pain following a period without pain lasting at least 4 weeks. Therefore pain flare-ups were registered no earlier than 4 weeks after the start of treatment, i.e. starting from Visit 5 (38 days after the start of treatment). The occurrence of pain flare-up was determined by the investigator.
  Percentages of patients with at least one pain flare-up resulting in consultancy with physician or professional management, resulting in disruption of daily activity, and resulting in NSAIDs intake were analyzed separately.
Time Frame: as for outcome 6
Population: Full Analysis Set (FAS). Denominator of proportion is the number of FAS patients who had at least one pain-free period and at least one pain flare-up episode during the study
Measure: Count of Participants; unit: Participants
Arm/Group | NSAIDs Group | NSAIDs+Milgamma+Milgamma Compositum Group
Number analyzed (Participants) | 35 | 10
Participants
  Patients with at least one pain flare-up resulting in consultancy with physician | 4 | 4
  Patients with at least one pain flare-up resulting in disruption of daily activity | 20 | 4
  Patients with at least one pain flare-up resulting in NSAIDs intake | 19 | 8
Statistical Analysis 1: Comparison: NSAIDs Group vs NSAIDs+Milgamma+Milgamma Compositum Group; Difference in proportion of patients with at least one pain flare-up resulting in consultancy with physician; Test type: Superiority; Difference in proportion = 28.6, 95% CI 2-sided [-3.6 to 60.7]
Statistical Analysis 2: Comparison: NSAIDs Group vs NSAIDs+Milgamma+Milgamma Compositum Group; Difference in proportion of patients with at least one pain flare-up resulting in disruption of daily activity; Test type: Superiority; Difference in proportion = -17.1, 95% CI 2-sided [-51.6 to 17.4]
Statistical Analysis 3: Comparison: NSAIDs Group vs NSAIDs+Milgamma+Milgamma Compositum Group; Difference in proportion of patients with at least one pain flare-up resulting in NSAIDs intake; Test type: Superiority; Difference in proportion = 25.7, 95% CI 2-sided [-4.1 to 55.5]

8. Secondary Outcome: Number of Treatment Days With NSAIDs
Description: Number of treatment days with NSAIDs was calculated using the data collected on the NSAIDs intake during the study irrespective of the specific drug used. Duration of each intake period was determined as Stop date - Start date +1 and, finally, all individual duration values were summed up. In case medication intake was ongoing at the End of Study Visit, stop date was imputed by the date of study completion.
Time Frame: From Baseline to Visit 9 (End of Study Visit, 94 days after the start of treatment)/ Early Discontinuation Visit
Population: Full Analysis Set (FAS)
Measure: Mean (Standard Deviation); unit: Days of treatment
Arm/Group | NSAIDs Group | NSAIDs+Milgamma+Milgamma Compositum Group
Number analyzed (Participants) | 244 | 250
Days of treatment | 9.6 (4.4) | 10.6 (8.9)
Statistical Analysis 1: Comparison: NSAIDs Group vs NSAIDs+Milgamma+Milgamma Compositum Group; NSAIDs intake during the study was analyzed. In order to calculate the total number of treatment days with NSAIDs, first, intersecting or adjacent records were collapsed, irrespective of the specific drug used; the duration of each of the resulting intake periods was determined as (End date - Start date + 1) and, finally, all individual duration values were summed up. In case medication intake was ongoing at the end of study, end date was imputed by the date of study completion; Test type: Superiority; p = 0.986, Wilcoxon (Mann-Whitney)

9. Secondary Outcome: Prescribed and Actual Number of Milgamma® Injections
Description: Prescribed number of Milgamma® injections was reported at Baseline visit. Actual number of injections was calculated by counting the number of injections administered and reported starting from Visit 2. If the treatment was interrupted, the days patient did not receive Milgamma® injections were not contribute to the total number of injections.
Time Frame: From Baseline to Visit 9 (End of Study Visit, 94 days after the start of treatment)/ Early Discontinuation Visit
Population: Safety population
Measure: Mean (Standard Deviation); unit: number of injections
Arm/Group | NSAIDs+Milgamma+Milgamma Compositum Group
Number analyzed (Participants) | 250
number of injections
  Prescribed exposure of Milgamma® injections | 9.3 (2.4)
  Actual exposure of Milgamma® injections | 9.3 (2.6)

10. Secondary Outcome: Prescribed and Actual Number of Treatment Days With Milgamma® Compositum
Description: Prescribed number of treatment days with Milgamma® compositum intake was reported at Baseline visit. Actual number of treatment days was calculated by summing up all the individual periods of treatment with Milgamma® compositum (in days) reported starting from Visit 2. If the treatment was interrupted, the days patient did not receive Milgamma® compositum were not contribute to the total number of treatment days with Milgamma® compositum intake.
Time Frame: From Baseline to Visit 9 (End of Study Visit, 94 days after the start of treatment)/ Early Discontinuation Visit
Population: Safety population
Measure: Mean (Standard Deviation); unit: Days of treatment
Arm/Group | NSAIDs+Milgamma+Milgamma Compositum Group
Number analyzed (Participants) | 250
Days of treatment
  Prescribed exposure of Milgamma® compositum | 30.1 (14.3)
  Actual exposure of Milgamma® compositum | 29.9 (13.2)

11. Secondary Outcome: Patient Satisfaction With Treatment
Description: Patient satisfaction with treatment was evaluated using a 5-point verbal rating scale (1= very dissatisfied, 2= dissatisfied, 3= neutral, 4= satisfied, 5= very satisfied) after 5, 10, 38 days and 3 months (94 days) since the start of treatment.
Time Frame: Visit 2 (5 days after the start of treatment); Visit 3 (10 days after the start of treatment); Visit 5 (38 days after the start of treatment) and Visit 9 (94 days after the start of treatment)
Population: Safety population
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | NSAIDs Group | NSAIDs+Milgamma+Milgamma Compositum Group
Number analyzed (Participants) | 244 | 250
units on a scale
  Visit 2 (5 days after the start of treatment) | 3.8 (0.8) | 3.8 (0.6)
  Visit 3 (10 days after the start of treatment) | 4.2 (0.8) | 4.1 (0.7)
  Visit 5 (38 days after the start of treatment) | 4.5 (0.7) | 4.5 (0.6)
  Visit 9 (94 days after the start of treatment) | 4.6 (0.6) | 4.7 (0.5)
Statistical Analysis 1: Comparison: NSAIDs Group vs NSAIDs+Milgamma+Milgamma Compositum Group; Comparison of patient satisfaction with treatment between treatment groups after 5 days since the start of study treatment; Test type: Superiority; p = 0.921, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: NSAIDs Group vs NSAIDs+Milgamma+Milgamma Compositum Group; Comparison of patient satisfaction with treatment between treatment groups after 10 days since the start of study treatment; Test type: Superiority; p = 0.051, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: NSAIDs Group vs NSAIDs+Milgamma+Milgamma Compositum Group; Comparison of patient satisfaction with treatment between treatment groups after 38 days since the start of study treatment; Test type: Superiority; p = 0.651, Wilcoxon (Mann-Whitney)
Statistical Analysis 4: Comparison: NSAIDs Group vs NSAIDs+Milgamma+Milgamma Compositum Group; Comparison of patient satisfaction with treatment between treatment groups after 3 months since the start of study treatment; Test type: Superiority; p = 0.106, Wilcoxon (Mann-Whitney)

12. Secondary Outcome: Percentage of Patients Prematurely Discontinued Milgamma®/ Milgamma® Compositum Treatment
Description: Percentage of patients prematurely discontinued prescribed treatment with Milgamma®/ Milgamma® compositum was evaluated by reasons for discontinuation.
Time Frame: From Baseline to Visit 9 (End of Study Visit, 94 days after the start of treatment)/ Early Discontinuation Visit
Population: Safety population
Measure: Count of Participants; unit: Participants
Arm/Group | NSAIDs+Milgamma+Milgamma Compositum Group
Number analyzed (Participants) | 250
Participants
  Completed prescribed step-therapy | 226
  Prematurely discontinued due to adverse event | 2
  Prematurely discontinued due to pain resolution | 19
  Prematurely discontinued due to patient's decision | 2
  Prematurely discontinued due to other reason | 1

13. Secondary Outcome: Reasons for Early Discontinuation of Study Participation
Description: Percentage of patient prematurely discontinued study participation by the following reasons: patient lost to follow-up, patient withdrew consent, administrative reasons, pain resolution, adverse event, death, other reason.
Time Frame: From Baseline to Visit 9 (End of Study Visit, 94 days after the start of treatment)/ Early Discontinuation Visit
Population: Safety population
Measure: Count of Participants; unit: Participants
Arm/Group | NSAIDs Group | NSAIDs+Milgamma+Milgamma Compositum Group
Number analyzed (Participants) | 244 | 250
Participants
  Patients completed the study in accordance with the protocol | 244 | 244
  Patients lost to follow-up | 0 | 0
  Patients withdrew informed consent | 0 | 1
  Patients discontinued study participation due to administrative reasons | 0 | 0
  Patients discontinued study participation due to pain resolution | 0 | 4
  Patients discontinued study participation due to adverse event | 0 | 0
  Patients discontinued study participation due to other reason | 0 | 1

14. Secondary Outcome: Frequency and Severity of Adverse Drug Reactions (ADRs)
Description: As this was a non-interventional study in which NSAIDs and Milgamma® / Milgamma® compositum were administered and managed within routine medical care, safety assessment was based on frequency and severity of Adverse Drug Reactions (ADRs) recorded during the study.
  ADR was defined as an adverse event (AE) suspected to be causally related to the medicinal product (Milgamma®, Milgamma® compositum or NSAID). The severity grade (mild, moderate or severe) of ADR was determined based on the investigator's judgement. Adverse events not related to the medicinal product were not monitored in this observational study.
Time Frame: From Baseline to Visit 9 (End of Study Visit, 94 days after the start of treatment)/ Early Discontinuation Visit
Population: Safety population was defined as all patients who signed informed consent for entry into the study and started the study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | NSAIDs Group | NSAIDs+Milgamma+Milgamma Compositum Group
Number analyzed (Participants) | 244 | 250
Participants
  Patients who had mild ADRs | 1 | 5
  Patients who had moderate ADRs | 0 | 0
  Patients who had severe ADRs | 0 | 0
  Patients who had not any ADRs | 243 | 245

ADVERSE EVENTS:
Time Frame: 3 months: from Baseline to Visit 9 (End of Study Visit, 94 days after the start of treatment)
Description: As this was a non-interventional study in which NSAIDs and Milgamma® / Milgamma® compositum were administered and managed within routine medical care, safety assessment was based on frequency and severity of Adverse Drug Reactions (ADRs) recorded during the study.
  ADR was defined as an adverse event (AE) suspected to be causally related to the medicinal product (Milgamma®, Milgamma® compositum or NSAID). Adverse events not related to the medicinal product were not monitored during this study.
Arm/Group | NSAIDs Group | NSAIDs+Milgamma+Milgamma Compositum Group
All-Cause Mortality (participants affected / at risk) | 0/244 | 0/250
Serious Adverse Events (participants affected / at risk) | 0/244 | 0/250
Other Adverse Events (participants affected / at risk) | 1/244 | 5/250
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NSAIDs Group (N=244) | NSAIDs+Milgamma+Milgamma Compositum Group (N=250)
ACNE (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
RASH ERYTHEMATOUS (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
URTICARIA (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
FACE OEDEMA (General disorders) | 0 (0) | 2 (2)
NAUSEA (Gastrointestinal disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2018-12-05): https://cdn.clinicaltrials.gov/large-docs/07/NCT03892707/Prot_000.pdf
  • Statistical Analysis Plan (2019-05-27): https://cdn.clinicaltrials.gov/large-docs/07/NCT03892707/SAP_001.pdf